CLINICAL TRIAL: NCT06571747
Title: Kaiser Permanente VACCination Improvement With Nudge-based CardiovAscular Targeted Engagement
Acronym: KP-VACCINATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: KP-VACCINATE
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases; Influenza; Behavior, Social
Keywords: Vaccination; Nudges; Behavioral Science; Cardiovascular Disease; Myocardial Infarction; Heart Failure; Implementation Science
MeSH Terms: conditions — Cardiovascular Diseases; Influenza, Human; Social Behavior; Myocardial Infarction; Heart Failure

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- CV Nudge/CV Nudge (Experimental): Intervention arms will test the effects of a cardiovascular-focused nudge communication developed using behavioral economic principles. This arm will receive the cardiovascular-focused nudge communication at 2 different timepoints during the influenza season.
  Interventions: Behavioral: Cardiovascular-Focused Nudge Communication
- CV Nudge/Usual Care (Experimental): Intervention arms will test the effects of a cardiovascular-focused nudge communication developed using behavioral economic principles. This arm will receive the cardiovascular-focused nudge communication at first timepoint and then usual care communication at the second timepoint during the influenza season.
  Interventions: Behavioral: Cardiovascular-Focused Nudge Communication
- Usual Care/CV Nudge (Experimental): Intervention arms will test the effects of a cardiovascular-focused nudge communication developed using behavioral economic principles. This arm will receive the usual care communication at first timepoint and then cardiovascular-focused nudge communication at the second timepoint during the influenza season.
  Interventions: Behavioral: Cardiovascular-Focused Nudge Communication
- Usual Care/Usual Care (No Intervention): The usual care arm will receive standard-of-care communication encouraging vaccination at both timepoints during the influenza season.

INTERVENTIONS:
Behavioral: Cardiovascular-Focused Nudge Communication — Intervention arms will receive a behavioral economic rooted nudge communication highlighting the potential cardiovascular benefits of vaccination.
  Arms: CV Nudge/CV Nudge; CV Nudge/Usual Care; Usual Care/CV Nudge

SUMMARY:
In randomized clinical trials and observational studies, influenza vaccination is effective in reducing influenza-related illness and hospitalizations and potentially cardiovascular (CV) events and mortality in select populations. However, the potential population-level benefit of influenza vaccination is limited by its uptake. Novel implementation strategies to improve vaccination uptake are needed.

KP VACCINATE is a multicenter, sequential, individual-level randomized controlled implementation trial examining the effectiveness of a CV-focused nudging communication vs. usual care communication on influenza vaccination uptake among Kaiser Permanente Northern California (KPNC) and Kaiser Permanente Mid Atlantic States (KPMAS) eligible members during the 2024-2025 influenza season.

DETAILED DESCRIPTION:
In randomized clinical trials and observational studies, influenza vaccination is effective in reducing influenza-related illness and hospitalizations and potentially cardiovascular events and mortality in select populations. However, the potential population level benefit of influenza vaccination is limited by its uptake. Novel implementation strategies to improve vaccination uptake are needed.

KP VACCINATE is a multicenter, sequential, individual-level randomized controlled implementation trial examining the effectiveness of a CV-focused nudging communication vs. usual care communication on influenza vaccination uptake among Kaiser Permanente Northern California (KPNC) and Kaiser Permanente Mid Atlantic States (KPMAS) eligible members during the 2024-2025 influenza season.

The study will evaluate an operational directive at KPNC and KPMAS. Eligible participants will be randomized into 4 study arms, corresponding to the messaging received at two different vaccine communication touchpoints (Touchpoint 1/Touchpoint 2) during the 2024-2025 influenza season:

1. CV-focused nudge communication/CV-focused nudge communication
2. CV-focused nudge communication/Usual care communication
3. Usual care communication/CV-focused nudge communication
4. Usual care communication/Usual care communication

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Active KPNC or KPMAS member
3. ≥6 months of continuous health plan coverage and prescription drug benefit before September 1, 2024
4. Evidence of member access to the KP HealthConnect® Portal and/or a listed registered email address
5. No documented influenza vaccination during the 2024-2025 influenza season prior to randomization

Exclusion Criteria:

1. Unable to receive or opted out of receiving health system messaging
2. Other exclusion that prevents messaging outreach.
3. Unknown service area or medical center affiliation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3668428 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with documented influenza vaccine receipt | up to 8 months
  Proportion of participants with documented influenza vaccine receipt after randomization.

SECONDARY OUTCOMES:
Time to influenza vaccine receipt | up to 8 months
  Time from randomization to influenza vaccine receipt.

OTHER OUTCOMES:
Laboratory-confirmed influenza infection | Up to 12 months
  Incidence of laboratory-confirmed influenza infection.
Hospitalization for influenza or pneumonia. | Up to 12 months
  Hospitalization for influenza or pneumonia.
All Cause Resource Utilization | Up to 12 months
  Composite and individual components of: All-cause hospitalization, emergency department (ED) visits, and observation stays
Total inpatient days | Up to 12 months
  Total inpatient days
All-cause intensive care unit (ICU) days | Up to 12 months
  All-cause intensive care unit (ICU) days
Major Adverse Cardiovascular Events | Up to 12 months
  Composite and individual components of major adverse CV events: incident or worsening heart failure events, hospitalization for acute myocardial infarction, atrial fibrillation, venous thromboembolism and hospitalization for acute stroke
All-cause death | Up to 12 months
  All-cause death, ascertained through a combination of Social Security Administration files, state death certificate files, electronic health records, and member proxy reporting.
Composite of major adverse CV events and all cause death | Up to 12 months
  Composite of major adverse CV events (incident or worsening heart failure events, hospitalization for acute myocardial infarction, atrial fibrillation, venous thromboembolism and hospitalization or acute stroke) and all-cause death.

CONTACTS AND LOCATIONS:
Overall Officials: Ankeet Bhatt, MD, Principal Investigator — The Permanente Medical Group; Benjamin Galper, MD, Principal Investigator — Mid-Atlantic Permanente Medical Group
Locations (2):
- United States (2):
  - Kaiser Permanente Northern California, Pleasanton, California
  - Kaiser Permanente Mid Atlantic States, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhatt AS, Berry NC, Parikh RV, Ballance Z, Tan TC, Marafino BJ, Hu H, Mummert M, Ambrosy AP, Hernandez-Diaz G, Fitch R, Patel S, Biering-Sorensen T, Claggett BL, Johansen ND, Jones A, Ku IA, Solomon SD, Vaduganathan M, Galper BZ, Lee KL, Go AS. Cardiovascular-Focused Messaging to Improve Influenza Vaccination Rates. NEJM Evid. 2025 Oct;4(10):EVIDoa2500208. doi: 10.1056/EVIDoa2500208. Epub 2025 Aug 30. PMID 40884406
- [Derived] Bhatt AS, Go AS, Parikh RV, Ballance Z, Tan TC, Marafino BJ, Hu H, Mummert M, Ambrosy AP, Hernandez-Diaz G, Fitch R, Patel S, Biering-Sorensen T, Claggett BL, Johansen ND, Jones A, Ku IA, Solomon SD, Vaduganathan M, Galper BZ, Lee KL, Berry NC; KP-VACCINATE Investigators. Electronically delivered, cardiovascular-focused messaging to improve influenza vaccination: Rationale, design, and baseline characteristics of the Kaiser Permanente VACCination Improvement with Nudge-based CardiovAscular Targeted Engagement (KP-VACCINATE) Megatrial. Am Heart J. 2025 Dec;290:129-139. doi: 10.1016/j.ahj.2025.06.007. Epub 2025 Jun 18. PMID 40541687